CLINICAL TRIAL: NCT06658379
Title: Prospective Validation Study of the CD8+TEMRA Cells As a Prognostic Biomarker of Healing Outcome After Fracture
Acronym: BioBone
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Unfallkrankenhaus Berlin (Other); Vivantes Klinikum Spandau (Unknown); University Hospital Dresden (Other); Universitaetsklinikum Muenster (Unknown); Leipzig University Hospital (Unknown); Jena University Hospital (Other); Beckman Coulter, Inc. (Industry); Federal Ministry of Education and Reserach (BMBF) (Unknown)
Responsible Party: Principal Investigator, Dr. Simon Reinke, Head of BIH Core Unit Cell and Tissue Harvesting, Charite University, Berlin, Germany
Other Study IDs: 01EK1514; DRKS00010872 (Other: german clinical trials register)
Record Dates: First submitted 2024-10-17; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Fracture Non Union; Fracture Healing; Long Bone Delayed-Union Fracture; Humerus Shaft Fracture; Forearm Fracture; Femoral Neck Fractures; Femur Distal Fracture; Pertrochanteric Fracture of Femur; Femoral Shaft Fracture; Proximal Tibia Fracture; Tibial Shaft Fracture; Distal Tibia Fracture
Keywords: long bone fracture; impaired fracture healing; fracture non-union; prognosis; prognostic biomarker; Immune system; T cells; radiology; bone fracture healing
MeSH Terms: conditions — Fractures, Ununited; Femoral Neck Fractures; Femoral Fractures, Distal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- fracture cohort: Humerus fracture, forearm fracture, femoral fracture. tibia fracture
  Interventions: Diagnostic Test: CD8+TEMRA

INTERVENTIONS:
Diagnostic Test: CD8+TEMRA

SUMMARY:
In approx. 10-15% of all fracture patients, there is a prolonged healing time or even a complete absence of fracture healing (non-union). As a result, these patients require further surgical interventions, combined with renewed or prolonged hospitalisation/rehabilitation and incapacity to work. To summarise, this therefore represents a serious socio-economic problem. At present, there is no prognostic method for the early prediction of patients at risk of a disturbed healing process. However, if these patients are successfully stratified, there are already a variety of therapeutic strategies available to additionally stimulate fracture healing. Therefore, the aim is to conduct a prospective clinical study to validate CD8+ TEMRA cells as a prognostic marker of impaired fracture healing. The investigators assume that preoperative CD8+ TEMRA cell expression represents a prognostic biomarker with high diagnostic precision for differentiating between a) normal healing patients, b) delayed healing patients and c) pseudarthrosis patients. Furthermore, the sensitivity and specificity should be high enough, health-economically significant and realisable in clinical routine.

DETAILED DESCRIPTION:
The aim is to identify high-risk patients before the initial operation based on their immunological profile and to be able to provide them with an improved, individualised therapeutic strategy. There are already a large number of approved therapeutic options that are currently only used in revision cases because, among other things, preoperative diagnostics and prognostics are lacking. Furthermore, a sufficient preoperatively determined biomarker would form the basis for the development of new therapeutic approaches, which represent a low cost-benefit and risk-benefit ratio.

The prospective biomarker validation study is applied in a routine-adapted procedure, i.e. all visits are part of the clinical radiological and functional routine checks. Blood sampling on arrival at the hospital will be used to determine the preoperative value of CD8+TEMRA cells. The healing process will be recorded using X-ray/CT images, radiological scores and functional clinical examinations as well as the SF-36. The 1st study endpoint (delayed healing) is after 17-19 weeks postoperatively, the 2nd study endpoint (pseudarthrosis) after 34-36 weeks. The validation of the biomarker will take place in a blinded procedure, whereby the predefined threshold value of the preoperative CD8+ TEMRA cell expression will be compared with the patient's healing status.

ELIGIBILITY:
Inclusion Criteria:

* male or female subjects
* subjects > 18 to 80 years of age at the time of screening
* closed fractures
* fractures of the humerus-shaft, forearm-shaft, femur and tibia
* Subjects suffering monotrauma or comparable with monotrauma, due to comparable post-surgery mobilisation
* osteosynthesis
* subject has signed an informed consent form
* legal capacity

Exclusion Criteria:

* cancer related fractures
* periprosthetic fractures
* known active Hepatitis B virus or Hepatitis C virus infection at screening
* known human immunodeficiency virus (HIV) infection, severe uncontrolled inflammatory disease or severe uncontrolled autoimmune disease (e.g., ulcerative colitis, Crohn's disease
* active malignancy or history of malignancy within 5 years prior to screening
* known diagnosis of moderate to severe dementia based on subject's medical history or severe psychiatric disorder
* known history of drug or alcohol abuse in the past 12 months, based on self-report or medical record
* history of autologous/allogeneic bone marrow (BM) or solid organ transplantation
* exposure to allogeneic cell-based therapy in the past or exposure to autologous cell therapy in the last 12 months before screening
* pregnancy
* subject is currently enrolled in an investigational device or drug trial, or has not yet completed a period of at least 30 days since ending other investigational device or drug trial(s).
* subject is detained or institutionalized under a court order or administrative order
* in the opinion of the investigator, the subject is unsuitable for participating in the study (patient compliance).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: University Hospital UniversityCentre for Orthopaedics and Trauma Surgery Dresden Charité Universitätsmedizin Berlin Centre for Musculoskeletal Surgery Clinic for Orthopaedics and Trauma Surgery Jena/Eisenberg Clinic Trauma Hospital Berlin Berlin Vivantes Hospital Spandau Berlin Clinic University Hospital Clinic and Polyclinic for Orthopaedics, Trauma Surgery and Plastic Surgery Leipzig
Sampling Method: Probability Sample
Enrollment: 640 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Clinical assessement of the fracture consolidation at first study endpoint based on radiological images | From surgery to 19 weeks post surgery
  Clinical assessement of the fracture consolidation (yes/no) based on radiological images at primary end point

SECONDARY OUTCOMES:
clinical assessement of the fracture consolidation at second study endpoint based on radiological images | From surgery to 36 weeks post surgery
  fracture consolidation (yes/no) after 36 weeks post surgery based on radiological images.

OTHER OUTCOMES:
Ability to work | From surgery to 1 year post surgery
  Period of return to work in days
Proportion of subjects with an additional intervention independent of a surgical or non-surgical treatment to foster the fracture healing process | From surgery to 1 year post surgery
  Number of surgically invasive and non-invasive measures
Duration of Physiotherapy | From surgery to 1 year post surgery
  Duration of physiotherapy sessions (units) done with a professional post-surgery.
Weight bearing and fracture healing | From surgery to 1 year post surgery
  Time to complete full weight bearing post surgery (weeks).
Rehabilitation and fracture healing | From surgery to 1 year post surgery
  Proportion of subjects with inpatient or day-care rehabilitation post surgery.
Infection rate | From surgery to 1 year post surgery
  Proportion of subjects with postoperative infections

CONTACTS AND LOCATIONS:
Overall Officials: Simon Reinke, Phd, Principal Investigator — Charité Universitätsmedizin Berlin, BIH Center for Regenerative Therapies (BCRT)
Locations (7):
- Germany (7):
  - Clinic for Trauma, Hand and Reconstructive Surgery University Hospital Münster (UKM), Münster, North Rhine-Westphalia
  - University Hospital University Centre for Orthopaedics and Trauma Surgery Dresden, Dresden, Saxony
  - University Hospital Clinic and Polyclinic for Orthopaedics, Trauma Surgery and Plastic Surgery Leipzig, Leipzig, Saxony
  - Unfallkrankenhaus Berlin, Berlin, State of Berlin
  - Charité Universitätsmedizin Berlin, Centre for Musculoskeletal Surgery (CMSC), Berlin, State of Berlin
  - Vivantes Klinikum Spandau Berlin, Berlin, State of Berlin
  - Clinic for Orthopaedics and Trauma Surgery Jena/Eisenberg, Eisenberg, Thuringia

IPD SHARING:
Plan to Share IPD: No
For data protection reasons, no individual participant data will be shared